CLINICAL TRIAL: NCT07045909
Title: A Phase 2, Open-label, Multicenter Multi-cohort Study to Evaluate the Efficacy and Safety of Anitocabtagene Autoleucel in Participants With Newly Diagnosed Multiple Myeloma
Brief Title: Efficacy and Safety of Anitocabtagene Autoleucel in Participants With Newly Diagnosed Multiple Myeloma (GEM-AnitoFIRST)
Acronym: GEM-AnitoFIRST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-AnitoFIRST
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: De Novo Multiple Myeloma; Anitocabtagene Autoleucel
MeSH Terms: interventions — daratumumab; isatuximab; Bortezomib; Lenalidomide; Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Phase 2, open-label, multicenter multicohort trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Experimental): Cohort A participants will be transplant eligible. Cohort A participants will receive induction with 6 cycles D-VRd. After induction, lymphodepleting chemotherapy will be administered consisting of cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day intravenous (IV) daily for 3 days before administration of anitocabtagene autoleucel. Initiation of the 3-day lymphodepleting chemotherapy regimen on Day -7 or Day -6 prior to the anitocabtagene autoleucel infusion on Day +1 is permitted. After lymphodepletion, participants will receive a single infusion of anitocabtagene autoleucel administered IV. After CAR T-cell infusion, cohort A participants will receive maintenance therapy with lenalidomide 10 mg daily for 2 years or until unacceptable toxicity, progression as per IMWG criteria, participant withdrawal of consent, death, or study completion, whichever occurs first.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anitocabtagene Autoleucel
- Cohort B (Experimental): Cohort B participants will not be transplant eligible. Cohort B participants will receive induction with 4 cycles Isa-VRd. After induction, lymphodepleting chemotherapy will be administered consisting of cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day IV daily for 3 days before administration of anitocabtagene autoleucel. Initiation of the 3-day lymphodepleting chemotherapy regimen on Day -7 or Day -6 prior to the anitocabtagene autoleucel infusion on Day +1 is permitted. After lymphodepletion, participants will receive a single infusion of anitocabtagene autoleucel administered IV. After CAR T-cell infusion, cohort B participants will receive maintenance therapy with lenalidomide 10 mg daily for 2 years or until unacceptable toxicity, progression as per IMWG criteria, participant withdrawal of consent, death, or study completion, whichever occurs first.
  Interventions: Drug: Isatuximab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anitocabtagene Autoleucel
- Cohort C (Experimental): Cohort C participants will not be transplant eligible. Cohort C participants will receive induction with 4 cycles Isa-VRd; 2 cycles followed by leukapheresis for T-cell collection to manufacture anitocabtagene autoleucel, followed by 2 additional cycles. After induction, lymphodepleting chemotherapy will be administered consisting of cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day IV daily for 3 days (Days -5 through -3) before administration of anitocabtagene autoleucel. The fludarabine dose may be adjusted for renal function. Initiation of the 3-day lymphodepleting chemotherapy regimen on Day -7 or Day -6 prior to the anitocabtagene autoleucel infusion on Day +1 is permitted. After lymphodepletion, participants will receive a single infusion of anitocabtagene autoleucel administered IV with a dose of 115 x 10e6 (± 10 x 10e6) CAR+ viable T cells. After CAR T-cell infusion, cohort C participants will not receive maintenance therapy.
  Interventions: Drug: Isatuximab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anitocabtagene Autoleucel

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered by subcutaneous (SC) injection.
  Arms: Cohort A
Drug: Isatuximab — Isatuximab will be administered IV.
  Arms: Cohort B; Cohort C
Drug: Bortezomib — Bortezomib dose will be calculated using the patient's actual body surface area at baseline and will be administered by SC injection.
Drug: Lenalidomide — Lenalidomide will be administered by oral route (all cohorts at induction, and cohorts A and B at maintenance).
Drug: Cyclophosphamide — As part of lymphodepleting therapy before CAR-T manufacture, administered IV.
Drug: Fludarabine — As part of lymphodepleting therapy before CAR-T manufacture, administered IV
Drug: Anitocabtagene Autoleucel — Single infusion IV

SUMMARY:
The goal of this clinical trial is to learn if anitocabtagene autoleucel following induction therapy works to treat adult participants with newly diagnosed multiple myeloma. The main objectives of this clinical trial are:

* To determine the incidence and severity of all adverse events (AEs).
* To determine the proportion of patients achieving undetectable minimal residual disease (uMRD) negative-CR rate (minimum 10 to -5) at 12 months (+/- 3 months) after enrollment.

Participants will receive induction therapy with a quadruplet regimen including a proteasome inhibitor (Bortezomib [V]), immunomodulatory drug (Lenalidomide [R]), dexamethasone [d] and anti-CD38 monoclonal antibody (Daratumumab [D] or Isatuximab [Isa]) followed by anitocabtagene autoleucel. Participants in Cohorts A and B will receive lenalidomide maintenance therapy following infusion with anitocabtagene autoleucel.

DETAILED DESCRIPTION:
Approximately 30 participants will be enrolled to receive induction therapy followed by a single dose of anitocabtagene autoleucel (~ 10 patients treated at target treatment dose per cohort). Participants will be distributed in 3 cohorts of treatment (A, B and C). Participants of cohort A will be transplant eligible while participants of cohorts B and C will not be planned to receive transplantation:

1. Induction therapy:

   * Cohort A: will consist of a total of 6 cycles D-VRd (28-day cycles); 3 cycles followed by leukapheresis for T-cell collection to manufacture anitocabtagene autoleucel, followed by 3 additional cycles.
   * Cohort B: will consist of a total of 4 cycles Isa-VRd (42-day cycles); 2 cycles followed by leukapheresis for T-cell collection to manufacture anitocabtagene autoleucel, followed by 2 additional cycles.
   * Cohort C: will consist of a total of 4 cycles Isa-VRd (42-day cycles); 2 cycles followed by leukapheresis for T-cell collection to manufacture anitocabtagene autoleucel, followed by 2 additional cycles.
2. Bridging Therapy:

   Bridging therapy will not be required because the leukapheresis and manufacturing will be planned during the induction phase to allow the availability of anitocabtagene autoleucel at the end of the induction therapy.
3. Lymphodepleting Chemotherapy:

   Chemotherapy regimen consisting of cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day will be administered intravenously (IV) daily for 3 days (Days -5 through -3) before administration of anitocabtagene autoleucel. The fludarabine dose may be adjusted for renal function. Initiation of the 3-day lymphodepleting chemotherapy regimen on Day -7 or Day -6 prior to the anitocabtagene autoleucel infusion on Day +1 is permitted.
4. Anitocabtagene Autoleucel:

   Treatment consists of a single infusion of anitocabtagene autoleucel administered intravenous (IV) on Day 1 at a target dose of 115 x 10e6 (± 10 x 10e6) CAR+ viable T cells.
5. Maintenance Therapy:

Cohorts A and B will receive maintenance therapy which will consist of lenalidomide 10 mg daily (days 1 to 28 of repeated 28-day cycle) for 2 years or until unacceptable toxicity, progression as per IMWG criteria, participant withdrawal of consent, death, or study completion, whichever occurs first. If any of these circumstances occur participant maintenance will end. After 3 cycles of lenalidomide maintenance, the dose can be increased to 15 mg orally once daily if tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Multiple Myeloma according to the IMWG criteria published in 2014.

   1. For cohort A, patients will ≤ 70 years of age.
   2. For the cohorts B and C, patients will be ≤ 80 years of age.
2. Measurable disease at screening per IMWG, defined as any of the following:

   1. Serum M-protein level ≥ 1 g/dL or urine M-protein level ≥ 200 mg/24 hours; or
   2. Light chain MM without measurable disease in the serum or urine: serum free light chain ≥ 10 mg/dL and abnormal serum free light chain ratio.

      * Note: Local laboratory results may be used to establish measurable disease at screening if the results are ≥ 125% of requirements.
3. Only participants who are candidates to receive either D-VRd or Isa-VRd induction regimens, as determined by the investigator, should be considered for this study.
4. Male or female aged 18 years or older and has capacity to give informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate hematological function defined as the following:

   * Hemoglobin count ≥ 7.5 g/dL (without any red blood cell [RBC] transfusion within 7 days prior to the test result; use of recombinant human erythropoietin is permitted).
   * Absolute neutrophil count (ANC) ≥ 500/μL (without non-PEGylated myeloid growth factor support within 7 days or PEGylated myeloid growth factor support within 14 days prior to the test result).
   * Platelet count ≥ 75,000/μL (unless secondary to bone marrow or spleen involvement of MM, in which platelet count ≥ 50,000/μL is permitted) without any platelet cell transfusion within 7 days prior to the test result. Bone marrow involvement by MM is demonstrated by bone marrow aspiration or biopsy. Spleen involvement by MM is demonstrated by splenomegaly.
   * Absolute lymphocyte count (ALC) ≥ 100/μL.
   * PTT/PT/INR < 1.5x upper limit of normal (ULN), unless on a stable dose of anticoagulant for a thromboembolic even (subjects with a history of thromboembolic stroke or history of Grade 2 or greater hemorrhage within 1 year are excluded.
7. Adequate renal, hepatic, pulmonary, and cardiac function defined as the following:

   * Estimated glomerular filtration rate (eGFR) (as estimated by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation [Section 12.14]) ≥ 45 mL/min.
   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   * Total bilirubin ≤ 1.5 mg/dL, except in participants with Gilbert's syndrome or documented MM liver or pancreatic involvement where ≤ 3 x ULN is permitted.
   * Cardiac ejection fraction ≥ 45% with no evidence of clinically significant pericardial effusion as determined by echocardiogram (ECHO). Multigated acquisition (MUGA) scan may be used if an ECHO is not available at the site.
   * No evidence of Grade 2 or higher (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0) pleural effusion or ascites (participants with Grade 1 pleural effusion or ascites are eligible).
   * Baseline oxygen saturation >92% on room air.
8. Females of childbearing potential must have a medically supervised negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential; refer to Section 12.2).
9. Willing to comply with and able to tolerate study procedures, including consent to participate in separate Long-term Safety Follow-up lasting up to 15 years per authorities´ guidance.

Exclusion Criteria:

1. Active or prior history of central nervous system (CNS) or meningeal involvement of MM.
2. Cardiac atrial or cardiac ventricular MM involvement.
3. Diagnosis of primary amyloidosis (AL), monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia (PCL), active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or Waldenstrom's macroglobulinemia at the time of screening.
4. Active malignancy (other than MM) requiring ongoing treatment for disease control within the last 24 months. Myelodysplastic syndrome (even without ongoing treatment) is not permitted. Allowed malignancy exceptions are:

   1. Localized skin cancer (melanoma and nonmelanoma) that has been completely resected and considered curative within the last 24 months is eligible.
   2. Cervix carcinoma in situ that has been completely resected and considered curative within the last 24 months is eligible.
   3. Bladder carcinoma in situ that has been completely resected and considered curative within the last 24 months is eligible.
   4. Breast carcinoma in situ that has been completely resected and considered curative within the last 24 months is eligible. Hormonal therapy after curative-intent treatment is permitted.
   5. Prostate cancer that is low grade and localized (Grade Group 1, has not spread to nearby lymph nodes [N0] or metastasized [M0]) within the last 24 months is eligible, including cases under surveillance only as part of standard of care. Androgen deprivation therapy is permitted.
   6. Localized renal cell carcinoma (≤ Stage 2) that has been completely resected and considered curative within the last 24 months is eligible.
   7. Localized (Stage 1) colorectal cancer that has been completely resected and considered curative (without need for adjuvant chemotherapy) within the last 24 months is eligible.
5. Any prior systemic anti-myeloma treatment (including BCMA-directed treatment) and/or radiotherapy before enrollment. Palliative radiation and corticosteroids (up to cumulative dose of 160mg prednisone or equivalent, and not requiring ongoing therapy) prior to enrollment are permitted. Participants must have recovered from all radiation-related toxicities. Patients with radiation-induced lung injury (RILI, radiation pneumonitis) during screening are excluded.
6. Prior allogeneic stem cell transplant (allo-SCT) (even if for another malignancy)
7. Live vaccine ≤ 4 weeks before enrollment and/or anticipating needing the vaccine during study period.
8. Presence or suspicion of fungal, bacterial, viral, or other infection that is systemic uncontrolled or requiring IV antimicrobials for management. Simple urinary tract infections and uncomplicated bacterial pharyngitis are permitted if the participant is responding to active treatment and satisfies the criteria of being afebrile (i.e., temperature < 38°C) for at least 24 hours prior to the investigator confirming the participant's eligibility.
9. Acute or chronic active hepatitis A, B, or C infection. Participants with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines or applicable country guidelines.
10. Human immunodeficiency virus (HIV)-seropositive.
11. Participants with history or presence of chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal will not be permitted to receive anti-CD38 monoclonal antibody in combination with VRd therapy; Note: FEV1 testing is required for participants who are planned
12. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months before enrollment.

    a. History or presence of intracranial or CNS disorder, such as hemorrhage, dementia, altered mental status, cerebellar disease, or any autoimmune disease with CNS involvement, PRES, or cerebral edema with confirmed structural defects by appropriate imaging. History of stroke or transient ischemic attack within 12 months before enrollment, or seizure disorders requiring active anticonvulsive medication. Patient with history of neurodegenerative disease (e.g., Parkinson's or Alzheimer's disease) must be excluded.
13. Peripheral neuropathy of Grade 3 or higher (per CTCAE v5.0; participants with Grade 2 peripheral neuropathy are eligible).
14. History of solitary plasmacytoma
15. History of autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in or requiring systemic immunosuppression or systemic disease-modifying agents within 2 years.
16. History of concomitant genetic syndrome associated with bone marrow failure, such as Fanconi anemia, Kostmann syndrome, or Shwachman-Diamond syndrome.
17. History of DVT or PE within 6 months before enrollment. Anticoagulants (e.g., warfarin, low-molecular weight heparin, Factor Xa inhibitors) are allowed if DVT/PE occurred > 6 months before enrollment, and if the participant is on a stable maintenance dose.
18. Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, G/J tube, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as Port-a-Cath or Hickman catheter are permitted.
19. Major surgery within 28 days before enrollment, or planned surgery required during study participation.
20. Any medical, neurologic or psychiatric condition that in the investigator's opinion is likely to interfere with study procedures including assessment of safety or efficacy of the study treatment.
21. Females who are pregnant or breastfeeding (due to the potentially dangerous effects of the lymphodepleting chemotherapy or induction regimen on the fetus or infant).
22. Participants of both sexes who are not willing to practice highly effective birth control from the time of consent through 12 months following lymphodepleting chemotherapy administration, 12 months after the completion of anitocabtagene autoleucel, 5 months after the last dose of isatuximab, 3 months after the last dose of daratumumab, bortezomib, or 28 days after the last dose of lenalidomide, whichever is longer (refer to Section 12.2). Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential. Participants of both sexes must also comply with any relevant REMS or aRMMs as part of an RMP. Additional information is in Section 6.3.1.
23. As per the investigator's judgment, the participant is unlikely to complete all protocol required study visits or procedures, including follow-up visits, or comply with or tolerate the study requirements for participation (e.g., participants who are at a risk for a thromboembolic event and are not willing to take venous thromboembolism prophylaxis should be excluded).
24. Contraindication to fludarabine or cyclophosphamide.
25. History of allergy or hypersensitivity to any study agent or study drug components. Participants with a history of severe hypersensitivity reaction to dimethyl sulfoxide (DMSO) are excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of all adverse events (AEs) | 3 years
  To characterize the safety of anitocabtagene autoleucel following induction therapy (incidence of treatment-emergent adverse events).
Undetectable minimal residual disease (uMRD) negative-CR rate (minimum 10-5) at 12 months (+/- 3 months) after enrollment. | 12 months
  To further characterize the efficacy profile of anitocabtagene autoleucel following induction therapy. MRD measured by Next Generation Flow Cytometry (NGF, with a sensitivity level of 10-6).

SECONDARY OUTCOMES:
Undetectable minimal residual disease (MRD) negative CR rate (minimum 10-5) at 2, 6, 12, 18 and 24 months after CAR T infusion and sustained undetectable minimal residual disease (uMRD) annually. | 2 years
  To further characterize the efficacy profile of anitocabtagene autoleucel following induction therapy. MRD measured by Next Generation Flow Cytometry.
Stringent complete response (sCR) or complete response (CR) rate, as assessed by investigators according to the International Myeloma Working Group (IMWG) criteria. | 6 months
  CR measured by cytomorphplogy and flow cytometry.
Overall MRD negativity (minimum 10e-5) | 3 years
  MRD measured by Next Generation Flow Cytometry.
Rate of conversion from undetectable to detectable MRD as well as biochemical progression rate. | 3 years
  MRD measured by Next Generation Flow Cytometry. Biochemical progression by measuring serum and/or urine monoclonal protein alone or with clinical features suggestive of progression including CRAB (C, hypercalcemia; R, renal failure; A, anemia; B, bone disease) symptoms.
Time to biochemical progression (including the conversion from undetectable to detectable MRD). | 3 years
  MRD measured by Next Generation Flow Cytometry. Serum and/or urine monoclonal protein alone or with clinical features suggestive of progression including CRAB (C, hypercalcemia; R, renal failure; A, anemia; B, bone disease) symptoms.
Undetectable MRD at 10e-6 (0.0001%) | 3 years
  MRD measured by Next Generation Flow Cytometry. Undetectable MRD at 10e-6 (10 elevated to -6, which is the same as 0.0001%) means no presence of multiple myloma cells within 1,000,000 cells analyzed by flow cytometry
Overall Response Rate (ORR) per International Myeloma Working Group (IMWG) criteria | 3 years
  ORR is defined as the proportion of participants who achieve a best overall response of at least partial response (PR) or better (sCR, CR, VGPR, or PR) per IMWG criteria.
Duration of Response (DoR) | 3 years
  DOR is derived only among participants who experience an overall response (sCR, CR, VGPR, or PR) per IMWG criteria and is defined as the time from first overall response to disease progression per IMWG criteria, or death from any cause, whichever occurs first.
Progression Free Survival (PFS) | 3 years
  PFS is defined as the time from enrollment to the first documented disease progression per IMWG criteria as determined by investigator assessed or death due to any cause, whichever occurs first.
Overall survival (OS) | 3 years
  OS is defined as the time from enrollment to the date of death from any cause.
Overall rate of "imaging plus MRD negative" (using PET/CT per International Myeloma Working Group [IMWG] criteria) | 3 years
  Measured by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan using the Deauville score.
  The Deauville score is a 5-point grading system used on FDG PET/CT imaging to assess treatment response. It is based on comparing FDG uptake in lesions with uptake in the liver and mediastinum. The Deauville score values are:
  1. No FDG uptake above background.
  2. Uptake less than the liver.
  3. Uptake equal to the liver.
  4. Uptake moderately greater than the liver.
  5. Uptake markedly greater than the liver, typically 2-3 times greater.
Expansion and persistence of anitocabtagene autoleucel in peripheral blood | 2.5 years
  Measured by Next Generation Flow Cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: María Victoria Mateos, MD PhD, Principal Investigator — Hospital Universitario de Salamanca (Salamanca); Jesús San Miguel, Professor, Study Director — Clínica Universidad de Navarra (Pamplona); Juan José Lahuerta, MD PhD, Study Chair — Hospital Universitario 12 de Octubre (Madrid); Joan Bladé, MD PhD, Study Chair — Hospital Clínic i Provincial de Barcelona (Barcelona)
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol (ICO BADALONA), Badalona
  - H. Clinic de Barcelona, Barcelona
  - H. 12 de Octubre, Madrid
  - H. Ramón y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario Salamanca, Salamanca
  - H. Marqués de Valdecilla, Santander
  - C H Santiago de Compostela, Santiago de Compostela
  - Complejo Hosp. Regional Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe de Valencia, Valencia